CLINICAL TRIAL: NCT01285596
Title: An Open-label, Randomized, 2-way Crossover Study to Evaluate the Pharmacokinetics of Mirabegron and Its Metabolites in Healthy Young and Elderly Male and Female Subjects
Brief Title: A Study to Evaluate How Mirabegron Enters and Leaves the Bloodstream According to Age and Sex
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 178-CL-072; 2008-006005-16 (EudraCT Number)
Record Dates: First submitted 2011-01-18; First posted 2011-01-28 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Healthy Volunteers; Pharmacokinetics of Mirabegron
Keywords: Pharmacokinetics; Cardiography; Impedance; Age groups; Gender Identity
MeSH Terms: interventions — mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Mirabegron — oral
  Other Names: YM178

SUMMARY:
Young and elderly, male and female subjects are each given 2 different doses of mirabegron for 7 days each. Levels of mirabegron in the blood are assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy elderly subject aged 55 years or more OR Healthy young subject aged 18 to 45 years, inclusive
* Male must agree to sexual abstinence and/or use a highly effective method of birth control from screening until 3 months after last dose of study medication
* Female subject must be of non-child bearing potential, i.e. post menopausal, surgically sterilized (e.g. tubal ligation), hysterectomy in medical history, or must practice an adequate non-hormonal contraceptive method to prevent pregnancies. Non-hormonal contraceptive methods are defined as:

  * Sexual abstinence from 1 month before admission until 3 months after discharge, OR
  * Subject's sexual partner has been surgically sterilized (since at least 3 months prior to the screening), OR
  * Subject is under two (2) of the following contraceptive methods: A) Diaphragm with spermicide; B)Intrauterine device; C)Sexual partner is using condoms in combination with a spermicidal creamDuring the study the subject is willing to use 1 of the 3 following contraceptive methods: diaphragm with spermicide, intrauterine device or partner is using condoms in combination with a spermicidal cream
* Body Mass Index between 18.5 and 30.0 kg/m2, inclusive

Exclusion Criteria:

* Known or suspected hypersensitivity to Mirabegron or any components of the formulation used
* Pregnant or breast feeding within 6 months before screening assessment
* Any of the liver function tests (i.e. ALT, AST and Alkaline phosphatase) above the upper limit of normal at repeated measurements
* Any clinically significant history of asthma, eczema, any other allergic condition or previous severe hypersensitivity to any drug (excluding non-active Hay-fever)
* Any clinically significant history of any other disease or disorder - gastrointestinal, cardiovascular, respiratory, renal, hepatic, neurological, dermatological, psychiatric or metabolic as judged by the investigator
* Any clinically significant abnormality following the investigator's review of the pre-study physical examination, ECG and clinical laboratory tests
* A hemoglobin value <13 g/dl (8.1 mmol/l) for males or <12 g/dl (7.5 mmol/l) for females OR a hematocrit value <40.0% for males or <37% for females OR a Red Blood Cell count <4.5 T/l (4500 mm3) for males or <3.8 T/l (3800 mm3) for females at screening and/or on the day of admission into the clinical unit
* Abnormal pulse and/or blood pressure measurements at the pre-study visit as follows: Pulse <40 or >90 bpm; mean systolic blood pressure >160 mmHg (elderly) or >140 mmHg (young); mean diastolic blood pressure >100 mmHg (elderly) or >90 mmHg (young), blood pressure measurements taken in triplicate after subject has been resting in supine position for 5 min; pulse will be measured automatically
* A marked baseline prolongation of QT/QTc interval after repeated measurements of >450 ms, a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias or torsades de pointes, structural heart disease, or a family history of Long QT Syndrome (LQTS)
* Use of any prescribed or OTC (over-the-counter) drugs (including vitamins, natural and herbal remedies, e.g. St. John's wort) in the 2 weeks prior to admission to the Clinical Unit, except for occasional use of paracetamol (up to 3 g/day)
* Regular use of any inducer of liver metabolism (e.g. barbiturates, rifampin) in the 3 months prior to admission to the Clinical Unit
* Any use of drugs of abuse within 3 months prior to admission to the Clinical Unit
* History of drinking more than 21 units of alcohol for males or more than 14 units of alcohol per week for females (1 unit = 270 cc of beer or 40 cc of spirits or 1 glass of wine) within 3 months prior to admission to the Clinical Unit
* Positive test for drugs of abuse or positive alcohol test at screening and/or on the day of admission into the clinical unit
* History of smoking more than 10 cigarettes (or equivalent amount of tobacco) per day within 3 months prior to admission to the Clinical Unit
* Participation in any clinical study within 3 months or participation in more than 3 clinical studies within 12 months, prior to the expected date of enrolment into the study
* Donation of blood or blood products within 3 months prior to admission to the Clinical Unit
* Positive serology test for HBsAg, anti HAV (IgM), anti-HCV or anti-HIV 1+2
* Subjects who, in the opinion of the investigator, are not likely to complete the trial for any reason
* Any clinical condition, which, in the opinion of the investigator would not allow safe completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2009-03; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Assessment of pharmacokinetics of mirabegron and its metabolites | Days 6 - 14 + Days 21 - 29

SECONDARY OUTCOMES:
Impedance cardiography assessed through evaluation of cardiac outputs, stroke volume, systemic vascular resistance index, mean arterial blood pressure and heart rate | Days -1, 1, 6 and 7

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Europe B.V.
Locations (1):
- Paris, France

REFERENCES:
- [Background] Krauwinkel W, van Dijk J, Schaddelee M, Eltink C, Meijer J, Strabach G, van Marle S, Kerbusch V, van Gelderen M. Pharmacokinetic properties of mirabegron, a beta3-adrenoceptor agonist: results from two phase I, randomized, multiple-dose studies in healthy young and elderly men and women. Clin Ther. 2012 Oct;34(10):2144-60. doi: 10.1016/j.clinthera.2012.09.010. PMID 23063375